CLINICAL TRIAL: NCT00412802
Title: Validation of Enoxaparin Dose Adaptation in Patients With Moderate Renal Failure Hospitalized for an Acute Coronary Syndrome, the VALIDE Study
Brief Title: Adaptation Dose of Enoxaparin in Moderate Renal Failure Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: French Cardiology Society (Other)
Responsible Party: Dr Anissa Bouzamondo, French Society of Cardiology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-01
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Acute Coronary Syndrome; Renal Failure
Keywords: enoxaparine; acute coronary syndrome; renal failure; dose adaptation
MeSH Terms: conditions — Acute Coronary Syndrome; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): dose adaptation of Enoxaparine at the renal deficient patients
  Interventions: Drug: dose adaptation of Enoxaparin
- 2 (Active Comparator): No dose adaptation of Enoxaparine at renal normal patients
  Interventions: Drug: normal injection of Enoxaparine

INTERVENTIONS:
Drug: dose adaptation of Enoxaparin — A same initial dose of 1 mg/kg will be administrated to all patients. According to creatinine clearance, the next doses (every 12 hours subcutaneously) will be adjusted with a 25% dose reduction if creatinine clearance is comprised between 30 and 50 ml/min.
  Arms: 1
Drug: normal injection of Enoxaparine — No dose adaptation of Enoxaparine
  Arms: 2

SUMMARY:
The objective of the VALIDE study is to validate that a 25% dose reduction of enoxaparine in patients with moderate renal failure (creatinine clearance between 30 and 50 ml/min) and hospitalized for an acute coronary syndrome provides at steady state a similar anti Xa level in plasma compared to that obtained in patients without renal failure and receiving the usual dose of 1 mg/kg subcutaneously every 12 hours. 140 per - protocol patients are planned to be included.

DETAILED DESCRIPTION:
Included patients will be those hospitalized for an acute coronary syndrome with indication of enoxaparin treatment. A same initial dose of 1 mg/kg will be administrated to all patients. According to creatinine clearance, the next doses (every 12 hours subcutaneously) will be adjusted with a 25% dose reduction if creatinine clearance is comprised between 30 and 50 ml/min. After the fourth dose, the anti-Xa plasma levels (main endpoint) will be measured at peak (between 3 and 5 hours after dose administration). Residual values of antiXa will also be measured before the fifth dose administration (secondary criteria).

The objective is to demonstrate a bio-equivalence of efficacy on the anti-Xa values obtained in patients with moderate rela failure compared with patients with creatinine clearance higher than 50 ml/min.

Thrombotic and bleeding events will be recorded during hospitalisation. 140 per-protocol evaluable consecutive patients will have to be obtained: 70 with creatinine clearance higher than 50 ml/min and 70 patients with creatinin clearance between 30 and 50 ml/min.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for acute coronary syndrome
* Indication of enoxaparin treatment
* Informed consent

Exclusion Criteria:

* Myocardial infarction with ST elevation
* Inclusion later than 12 hours after the first enoxaparin dose administration
* Creatinine clearance lower than 30 ml/min
* History of thrombopenia induced by heparin
* Platelet count lower than 100.000 / mm3
* Age < 18
* Pregnancy
* History of hemorrhagic stroke
* Contra-indication to enoxaparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
plasma antiXa levels at peak after the fourth enoxaparine dose administration

SECONDARY OUTCOMES:
residual plasma antiXa level before the fifth enoxaparine dose administration
activated thromboplastin time
thrombotic events
bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Imad ABI NASR, MD, Study Chair — Ambroise Paré Hospital
Locations (9):
- France (9):
  - Sud Francilien Hospital center, Corbeil, Essonnes
  - CHU Jean MINJOZ, Besançon
  - Ambroise Paré Hospital, Boulogne
  - Henri Mondor Hospital, Créteil
  - Lagny center Hospital, Lagny-sur-Marne
  - Pitié Salpêtrière Hospital, Paris
  - CHU Bichat, Paris
  - Lariboisiére Hospital, Paris
  - Rangueil Hospital, Toulouse